CLINICAL TRIAL: NCT05454111
Title: A Randomized Control Trial to Compare the Efficacy and Safety of CARTO-Finder-guided Ablation Plus Pulmonary Vein Isolation and Multiscale Entropy-guided Ablation Plus Pulmonary Vein Isolation in Patients With Persistent Atrial Fibrillation
Brief Title: CARTO-Finder Guided Ablation Versus Multiscale Entropy Guided Ablation in Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Shandong University of Traditional Chinese Medicine (Other); Department of Cardiology, Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine (Unknown); Wuhan Central Hospital (Other); Jining Medical University (Other); Department of Cardiology, Yuhuan Second People's Hospital (Unknown); Department of Cardiology, Changshu Hospital of Traditional Chinese Medicine (Unknown); Department of Cardiology, The PLA Navy Anqing Hospital (Unknown); Department of Cardiology, Jinan City People's Hospital (Unknown); Department of Cardiology, Xuzhou Central Hospital (Unknown)
Responsible Party: Principal Investigator, Xu Liu, Professor, deputy director of cardiology department of Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Find-AF
Record Dates: First submitted 2022-07-05; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; catheter ablation; CARTO-Finder-guided ablation; Multiscale entropy-guided ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CARTO-Finder-guided ablation plus PVI (Active Comparator): Pulmonary vein circumferential isolation + + ablation of sites recognized by CARTO-Finder module as the core of rotors.
  Interventions: Procedure: CARTO-Finder-guided ablation plus PVI
- Multiscale entropy-guided ablation plus PVI (Experimental): Pulmonary vein circumferential isolation + ablation of sites recognized by multiscale entropy analysis as the core of rotors.
  Interventions: Procedure: Multiscale entropy-guided ablation plus PVI

INTERVENTIONS:
Procedure: Multiscale entropy-guided ablation plus PVI — The multiscale entropy is calculated based on intracardiac electrical signals, higher multiscale entropy value indicates closer to the core of rotors which maintains the persistent atrial fibrillation.
  Arms: Multiscale entropy-guided ablation plus PVI
Procedure: CARTO-Finder-guided ablation plus PVI — CARTO-Finder-guided ablation plus PVI
  Arms: CARTO-Finder-guided ablation plus PVI

SUMMARY:
This is a randomized control trial to compare the efficacy and safety of CARTO-Finder-guided ablation plus pulmonary vein isolation versus multiscale entropy (MSE)-guided pulmonary vein isolation in patients with persistent atrial fibrillation.

DETAILED DESCRIPTION:
This is a randomized control trial. Patients with persistent atrial fibrillation are enrolled and randomized to CARTO-Finder-guided ablation plus PVI group or MSE-guided ablation plus PVI group. Postoperative recurrence rate and other indicators are analyzed to compare the efficacy and safety between CARTO-Finder-guided ablation plus PVI and MSE-guided ablation plus PVI in patients with persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old
2. Persistent AF
3. Nonresponse or intolerance to ≥1 antiarrhythmic drug

Exclusion Criteria:

1. With uncontrolled congestive heart failure;
2. Having significant valvular disease;
3. Having moderate-to-severe pulmonary hypertension;
4. With myocardial infarction or stroke within 6 months of screening;
5. With Significant congenital heart disease;
6. Ejection fraction was <40% measured by echocardiography;
7. Allergic to contrast media;
8. Contraindication to anticoagulation medications;
9. Severe pulmonary disease e.g. restrictive pulmonary disease, chronic obstructive disease (COPD);
10. Left atrial thrombus;
11. Having any contraindication to right or left sided heart catheterization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation (AF)/atrial flutter (AFL)/atrial tachycardia (AT) recurrence rate | up to 24 months after enrollment
  AF/AFL/AT recurrence is defined as presence of documented AF/AFL/AT episodes of 30 seconds or longer duration

SECONDARY OUTCOMES:
Postoperative AF recurrence rate | up to 24 months after enrollment
  AF recurrence is defined as presence of documented AF episodes of 30 seconds or longer duration
Postoperative AFL/AT rate | up to 24 months after enrollment
  Occurrence of AFL/AT is defined as presence of documented AFL/AT episodes of 30 seconds or longer duration

OTHER OUTCOMES:
Changes in the diameter of the left atrium | up to 24 months after enrollment
  Changes in the diameter of the left atrium
Changes in the diameter of the left ventricular ejection fraction | up to 24 months after enrollment
  Changes in the diameter of the left ventricular ejection fraction
Incidence of complications | up to 24 months after enrollment
  death, atrio-esophageal fistula, cardiac tamponade/perforation, myocardial infarction, stroke/cerebrovascular accident, thromboembolism, diaphragmatic paralysis, pneumothorax, pleural effusion, heart block, pulmonary vein stenosis, pulmonary edema, left atrial thrombus, pericarditis and major vascular access complication or bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided